CLINICAL TRIAL: NCT01733446
Title: A Study of the Effect of Arterial Carbon Dioxide Tension on the Recovery of Spontaneous Respiration With Respiratory Inductance Plethysmography (RIP) During High Frequency Jet Ventilation (HFJV) Under General Anesthesia
Brief Title: A Study of the Effect of Arterial Carbon Dioxide Tension on the Recovery of Spontaneous Respiration
Acronym: RIP03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 816280
Record Dates: First submitted 2012-10-02; First posted 2012-11-27 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Surgery; Anesthesia
Keywords: High frequency jet ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard anesthesia regimen (No Intervention): Positive pressure ventilation will be stopped at the same time infusions of anesthetic agents and spontaneous ventilation employed until emergence from anesthesia is observed. (This is standard protocol for everyday anesthesia management of this population.)
- Continuation of High Frequency Jet Ventilation ( HFJV) (Experimental): In Group B after cessation of anesthetic infusions, High Frequency Jet Ventilation (HFJV) will continue through the endotracheal tube. Patient will be extubated when awake. Respiratory Inductance Plethysmography (RIP) and transcutaneous carbon dioxide (PtcCO2) measurements will continue for the duration of emergence.
  Interventions: Other: Continuation of High Frequency Jet Ventilation (HFJV)

INTERVENTIONS:
Other: Continuation of High Frequency Jet Ventilation (HFJV) — In Group B, after cessation of anesthetic infusions, High Frequency Jet Ventilation (HFJV) will continue through the endotracheal tube. Patient will be extubated when awake. Respiratory Inductance Plethysmography (RIP) and Transcutaneous carbon dioxide (PtcCO2) measurements will continue for the duration of emergence.
  Arms: Continuation of High Frequency Jet Ventilation ( HFJV)

SUMMARY:
The investigators data reveal an important new observation regarding the recovery of breathing during emergence from general anesthesia: respiration resumes as a prolonged abdominal expiration event.

The present study aims to further clarify the physiology of recovery of breathing with the addition of a cutaneous monitor for arterial carbon dioxide measurement and a comparison of two different recovery paradigms.

DETAILED DESCRIPTION:
The present study will use non-invasive respiratory inductance plethysmography(RIP) and transcutaneous carbon dioxide measurement to compare recovery of respiration under constant Transcutaneous carbon dioxide measurement( ptcCO2) with continuous high frequency jet ventilation HFJV (study method) with recovery of respiration during rising and apnea (current standard).

The investigators hypothesize that the prolonged abdominal expiration that we observed during recovery of breathing in prior studies will be unaffected by arterial carbon dioxide (CO2) levels.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female patients ages > 18 to < 80
2. Scheduled for procedures under general anesthesia with jet ventilation
3. Sign informed consent
4. Candidate for total intravenous anesthesia with propofol and remifentanil (which is standard protocol in this type of population)

Exclusion Criteria:

1. Absence of informed consent
2. No planned use intra-operative use of jet ventilation
3. Known difficulties with jet ventilation during prior surgical procedures
4. Emergency surgery
5. Baseline (oxygen saturation)SpO2 <92% on room air
6. BMI > 50
7. Pregnant or lactating females
8. Skin damage, rash or significant lesions in the areas covered by the RIP bands or transcutaneous CO2 sensor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-09; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
spontaneous breathing | Day 0 in the operating room occurring in the specific time frame of the end of anesthesia to patient 's first breath
  The primary variable will be first breath as detected by Respiratory Inductance Plethysmography (RIP. This will occur in the operating room at the end of the surgery and anesthesia.)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua H Atkins, MD PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States